CLINICAL TRIAL: NCT03803280
Title: Implementation of the Enhanced Recovery in Abdominal Surgery Pathway in the National Health Network (IMPRICA Project)
Brief Title: Implementation of Enhanced Recovery Protocol in Spain
Acronym: IMPRICA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grupo Español de Rehabilitación Multimodal (Other)
Collaborators: Instituto de Investigación Sanitaria Aragón (Other); Instituto Aragones de Ciencias de la Salud (Other Government)
Responsible Party: Sponsor
Other Study IDs: GERM03
Record Dates: First submitted 2019-01-11; First posted 2019-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Major Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional care: Patients with major abdominal surgery without before a enhanced recovery program was stablished
- ERAS care: Patients with major abdominal surgery within a enhanced recovery program was stablished
  Interventions: Procedure: ERAS program

INTERVENTIONS:
Procedure: ERAS program — ERAS pathway according to the Spanish Via RICA
  Groups: ERAS care

SUMMARY:
The main objective is the multicenter and uniform implementation of a agreed upon perioperative evidence based program emanated from the Enhanced Recovery for abdominal surgery pathway (RICA) published by the Spanish National Health Service and the Aragon Institute of Health, in hospitals of the National Health Network.

The evaluation and outcomes of such implementation is proposed as a secondary objective. Different established indicator will compared traditional care results with those from the new program in the short and medium term. 10 interested hospital centers are selected. In each of them a retrospective study will be conducted to analyze the clinical results obtained in abdominal surgery in the past six months. After making the necessary training to clinical teams and assure the project development and implementation in each center, a prospective study in which all patients in the program are being recruited will be held. Hospital stay as well as perioperative mortality and morbidity will be collected. We will analyze data from: days of hospital stay (potential and actual), efficiency (cost/procedure), quality of care, time to complete reintegration into family, social and labor environment and quality of life.

DETAILED DESCRIPTION:
A uniform, consensual and multicentric implementation of the multidisciplinary Perioperative Medicine Program is proposed, the program comes form the Clinical Pathway of Intensified Recovery in Abdominal Surgery -RICA-, published by the Spanish National Health System as clinical guideline.

It covers the perioperative area in complex abdominal surgery and extends from the moment of diagnosis in the Surgery office until the last revision performed one year after surgery.

It is proposed as a double study; a first retrospective analysis of the results and perioperative complications referred and available in the Centers involved in the study; and a second analysis of results after the implementation of the Program, in the same Centers. Once both are finished, the comparison between them and their communication will be carried out using the appropriate reports.

Actors: Multidisciplinary teams made up of nurses, surgeons, anesthesiologists, nutritionists / endocrinologists, physiotherapists and rehabilitators.

Patients: All patients recruited in the different hospitals for the RICA Perioperative Medicine Program susceptible to performing complex abdominal surgery.

Variables under study: Perioperative complications according to the Clavien-Dindo classification and the European Perioperative Clinical Outcome definitions (EPCO); Times of global hospital stay and in critical care units; the rate of readmissions and the complications derived from them, the rate of surgical reoperations, the analysis of cost per process (including the total cost in the study period-two years-), the time until complete reincorporation into the family environment and socio-labor, the indices of quality perceived by the patient and / or their caregivers, the final quality of life index obtained by each patient (resulting quality of life).

Data collection and analysis: Record of described variables were be included in an "on line"database available to all centers.

Limitations of the Study: impossibility to include all the patients that can be recruited in surgery consultations due to rejection of the staff (negative to the benchmarking and / or to the program) or negative of the patient. Loss of data in follow-up due to the failure of patients. Difficulty in analyzing costs due to lack of economic data in the Centers. Lack of motivation in the multidisciplinary teams. Rupture of the program in case of emergency / emergency.

Material and Methodology:

Participating Centers: Previously selected for their well-known Organizational capacity and their experience and interest.

First Phase: Realization of retrospective study of existing results in each Center in the six months prior to the implementation of the Program and Conformation of the multidisciplinary teams that will implement the Intensified Recovery Program.

Second phase: Training of the Teams in IACS (Instituto Aragones Ciencias de la Salud) on the implementation of enhanced recovery programs provided with online training through platform built "ad hoc" and in person for training with experts. Development of the Normalized Work Protocol (NTP) in each assigned Center and implementation of the forms and database in the Clinical History of the Centers (considering electronic Clinical History).

Third phase: Progressive recruitment of patients and inclusion in the Program (on-line database) and start of the one-year prospective study from the patient's inclusion.

Inclusion Criteria:

-Patients over 18 years old, scheduled for major abdominal surgical surgery, due to malignant or benign causes. (It is defined as complex major surgery that lasts more than two hours, it is estimated that it may require the transfusion of at least 2 red cell concentrates or it is estimated a loss greater than or equal to 15% of the patient's blood volumen).

ELIGIBILITY:
Inclusion Criteria:

• Patients over 18 years old, scheduled for major abdominal surgical surgery, due to malignant or benign causes.

Exclusion Criteria:

* Urgent Surgery.
* Patients ASA (American Society of Anesthesiology) IV or higher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old, scheduled for major abdominal surgical surgery, due to malignant or benign causes (It is defined as complex major surgery that lasts more than two hours or it is estimated that it may require the transfusion of at least 2 red cell concentrates or it is estimated a loss greater than or equal to 15% of the patient's blood volumen).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-07-15 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with postoperative complications | 30 days after surgery
  complications after surgery
Mortality | 3 years
  Number of patients dead after surgery
Long term mortality | 5 years
  Number of patients dead after surgery

SECONDARY OUTCOMES:
Hospital stay | perioperative stay
  Days of stay in hospital after surgery
compliance of the protocol | 1 month after surgery
  Rate of compliance of each ERAS (Enhanced Recovery After Surgery) item
re-admission | 1 month after surgery
  patient needing hospital stay after being at home after primary surgery
Cost | 1 month after surgery
  Price of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Calvo, Dr, Study Chair — Grupo Español de Rehabilitación Multimodal
Locations (3):
- Spain (3):
  - Hospital Universitario Infanta Leonor, Madrid
  - Complejo Hospitalario de Salamanca, Salamanca
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vorwald P, Bruna Esteban M, Ortega Lucea S, Ramirez Rodriguez JM; Grupo de Trabajo de Cirugia Esofagogastrica del Grupo Espanol de Rehabilitacion Multimodal (GERM). Enhanced recovery after esophageal resection. Cir Esp (Engl Ed). 2018 Aug-Sep;96(7):401-409. doi: 10.1016/j.ciresp.2018.02.010. Epub 2018 Mar 21. English, Spanish. PMID 29573788
- [Result] Bruna M, Navarro C, Baez C, Ramirez JM, Ortiz MA. Results of a national survey about perioperative care in gastric resection surgery. Cir Esp (Engl Ed). 2018 Aug-Sep;96(7):410-418. doi: 10.1016/j.ciresp.2018.03.004. Epub 2018 Apr 24. English, Spanish. PMID 29699695
- [Result] Ruiz-Tovar J, Munoz JL, Royo P, Duran M, Redondo E, Ramirez JM; Grupo Espanol de Rehabilitacion Multimodal (GERM). Implementation of the Spanish ERAS program in bariatric surgery. Minim Invasive Ther Allied Technol. 2018 Dec;27(6):365-372. doi: 10.1080/13645706.2018.1446988. Epub 2018 Mar 8. PMID 29519184
- [Result] Bruna Esteban M, Vorwald P, Ortega Lucea S, Ramirez Rodriguez JM; Grupo de Trabajo de Cirugia Esofagogastrica del Grupo Espanol de Rehabilitacion Multimodal (GERM). Enhanced recovery after surgery in gastric resections. Cir Esp. 2017 Feb;95(2):73-82. doi: 10.1016/j.ciresp.2016.10.013. Epub 2017 Feb 6. English, Spanish. PMID 28185641
- [Result] Martinez AB, Longas J, Ramirez JM. A model for lymphocyte activation in open versus laparoscopic surgery in colorectal cancer patients in enhanced recovery after surgery (ERAS) protocols. Int J Colorectal Dis. 2017 Jun;32(6):913-916. doi: 10.1007/s00384-016-2731-2. Epub 2016 Nov 30. PMID 27900463
- [Result] Ruiz-Tovar J, Royo P, Munoz JL, Duran M, Redondo E, Ramirez JM; GERM. Implementation of the Spanish National Enhanced Recovery Program (ERAS) in Bariatric Surgery: A Pilot Study. Surg Laparosc Endosc Percutan Tech. 2016 Dec;26(6):439-443. doi: 10.1097/SLE.0000000000000323. PMID 27753710
- [Result] Moya P, Soriano-Irigaray L, Ramirez JM, Garcea A, Blasco O, Blanco FJ, Brugiotti C, Miranda E, Arroyo A. Perioperative Standard Oral Nutrition Supplements Versus Immunonutrition in Patients Undergoing Colorectal Resection in an Enhanced Recovery (ERAS) Protocol: A Multicenter Randomized Clinical Trial (SONVI Study). Medicine (Baltimore). 2016 May;95(21):e3704. doi: 10.1097/MD.0000000000003704. PMID 27227930
- [Result] Gonzalez-Ayora S, Pastor C, Guadalajara H, Ramirez JM, Royo P, Redondo E, Arroyo A, Moya P, Garcia-Olmo D. Enhanced recovery care after colorectal surgery in elderly patients. Compliance and outcomes of a multicenter study from the Spanish working group on ERAS. Int J Colorectal Dis. 2016 Sep;31(9):1625-31. doi: 10.1007/s00384-016-2621-7. Epub 2016 Jul 4. PMID 27378580
- [Result] Esteban F, Cerdan FJ, Garcia-Alonso M, Sanz-Lopez R, Arroyo A, Ramirez JM, Moreno C, Morales R, Navarro A, Fuentes M. A multicentre comparison of a fast track or conventional postoperative protocol following laparoscopic or open elective surgery for colorectal cancer surgery. Colorectal Dis. 2014 Feb;16(2):134-40. doi: 10.1111/codi.12472. PMID 24164975
- [Result] Nygren J, Thacker J, Carli F, Fearon KC, Norderval S, Lobo DN, Ljungqvist O, Soop M, Ramirez J; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective rectal/pelvic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):285-305. doi: 10.1007/s00268-012-1787-6. No abstract available. PMID 23052796
- [Result] Arroyo A, Ramirez JM, Callejo D, Vinas X, Maeso S, Cabezali R, Miranda E; Spanish Working Group in Fast Track Surgery (GERM). Influence of size and complexity of the hospitals in an enhanced recovery programme for colorectal resection. Int J Colorectal Dis. 2012 Dec;27(12):1637-44. doi: 10.1007/s00384-012-1497-4. Epub 2012 May 27. PMID 22645075
- [Result] Ramirez JM, Blasco JA, Roig JV, Maeso-Martinez S, Casal JE, Esteban F, Lic DC; Spanish working group on fast track surgery. Enhanced recovery in colorectal surgery: a multicentre study. BMC Surg. 2011 Apr 14;11:9. doi: 10.1186/1471-2482-11-9. PMID 21489315